CLINICAL TRIAL: NCT04948775
Title: Effect of Cervical Stabilization Exercises on Cervical Proprioception, Functional Status and Quality of Life in Patients With Rheumatoid Arthritis
Brief Title: Cervical Stabilization Exercises in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Deniz Bayraktar, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RACSE
Record Dates: First submitted 2021-06-28; First posted 2021-07-02 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Proprioception; Exercise; Neck; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Cervical Stabilization Exercise Group
  Interventions: Other: Cervical stabilization exercises
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Other: Cervical stabilization exercises — A progressive home-based cervical stabilization exercise program which is aimed to train deep stabilizer muscles of the cervical spine and improve coordination between superficial and deep cervical muscles will be performed by the patients for 6 weeks. Exercises are going to be delivered by sending messages and video instructions via a freeware and crossplatform messaging service (WhatsApp Messenger) in a weekly basis.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to investigate the effectiveness of cervical stabilization exercises on cervical positioning error in rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, recurrent polyarthritis of the synovial joints. Although the prevalence of the disease shows ethnic differences, the average prevelance of the disease is 1%, and the female/male ratio is 2.5-3/1. The average age of onset is between 30-50 years. Common cervical involvement in RA patients was first described by Garrod in 1890. The most common inflammatory arthritis involving the cervical vertebra is RA. Thoracic and lumbar spine involvement is less common compared to cervical spine involvement in the disease.

Proprioceptive sense is defined as a type of specialized sensory model that includes joint movement (kinesthesia) and position sense. Mechanoreceptors located in different structures such as muscle, tendon, joint capsule and skin in both axial joints and peripheral joints provide the perception of joint position and movement. The sense of proprioception provides dynamic joint stability and various movement skills without the need for conscious planning. It also prevents premature joint degeneration by preventing uncontrolled load on the joints. The cervical proprioceptive system consists of mechanoreceptors of the cervical intervertebral joints, neck muscles and vertebral ligaments, muscle spindles localized in the deep muscles of the cervical spine, and sensitive fibers connecting the neurons in posterior horn of the spinal cord to the neck proprioceptors. Cervical vertebrae, unlike the thoracic and lumbar regions, has an additional importance due to the abundance of mechanoreceptors that provide reflex connections and proprioceptive input with the vestibular central and central nervous systems. In previous studies, it has been shown that the sense of cervical proprioception is impaired in patients with chronic neck pain due to traumatic and degenerative causes. It has been shown that cervical proprioceptive sensory dysfunction in RA causes, vestibular symptoms, changes in contol of eye movements and postural disorders in cervical paravertebral muscles.

No study investigating the effect of exercise on cervical proprioception in RA patients was found in the literature. The aim of this study was to determine the effects of cervical stabilization exercises on cervical proprioception in RA patients. The secondary aim of the present study is to evaluate the effects of cervical stabilization exercises on the functional status and quality of life in patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with RA according to the ACR 2010 Criteria
* Being between 18 and 65 years old
* To be able to understand the given commands

Exclusion Criteria:

* Refusing to participate in the study
* History of trauma involving the neck
* Having an orthopedic disorder concerning the neck
* History of spine surgery
* Having a disease that affects vestibular system
* Upper extremity involvement due to a disorder other than RA
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Reposition Error | At baseline and 6 weeks later
  Cervical reposition error method will be used to determine the cervical proprioception accuracy. Cervical reposition error will be evaluated in flexion, extension, rotation and lateral flexion directions and will be calculated using a special formula.

SECONDARY OUTCOMES:
Change in Functional Status | At baseline and 6 weeks later
  Neck Disability Index, which is a self-report tool and has 10 items, will be used to evalutae the functional status of the neck.
Change in Physical Performance | At baseline and 6 weeks later
  Neck flexor muscles endurance test and neck extansor muscles endurance test will be used to investigate physical performance.
Change in Disease Related Quality of Life | At baseline and 6 week later
  RAQoL (30 items, self-report) and HAQ (20 items, self-report) will be employed to evaluate the disease related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bayraktar, PT, PhD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon a reasonable request.
Time Frame: Data will be available from September 2023 to December 2043.
Access Criteria: Data will be send for academical purposes (for conducting a meta-analysis and/or systematic review)

REFERENCES:
- [Background] Harris ED Jr. Rheumatoid arthritis. Pathophysiology and implications for therapy. N Engl J Med. 1990 May 3;322(18):1277-89. doi: 10.1056/NEJM199005033221805. No abstract available. PMID 2271017
- [Background] Gillick JL, Wainwright J, Das K. Rheumatoid Arthritis and the Cervical Spine: A Review on the Role of Surgery. Int J Rheumatol. 2015;2015:252456. doi: 10.1155/2015/252456. Epub 2015 Aug 17. PMID 26351458
- [Background] Heywood AW, Meyers OL. Rheumatoid arthritis of the thoracic and lumbar spine. J Bone Joint Surg Br. 1986 May;68(3):362-8. doi: 10.1302/0301-620X.68B3.3733796.
- [Background] Roijezon U, Clark NC, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 1: Basic science and principles of assessment and clinical interventions. Man Ther. 2015 Jun;20(3):368-77. doi: 10.1016/j.math.2015.01.008. Epub 2015 Jan 29. PMID 25703454
- [Background] Armstrong B, McNair P, Taylor D. Head and neck position sense. Sports Med. 2008;38(2):101-17. doi: 10.2165/00007256-200838020-00002. PMID 18201114
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control--Part 2: case studies. Man Ther. 2008 Jun;13(3):266-75. doi: 10.1016/j.math.2007.11.002. Epub 2008 Jan 3. PMID 18180194
- [Derived] Gulcemal MO, Sarac DC, Alp G, Duran G, Gucenmez S, Solmaz D, Akar S, Bayraktar D. Effects of video-based cervical stabilization home exercises in patients with rheumatoid arthritis: a randomized controlled pilot study. Z Rheumatol. 2024 Dec;83(Suppl 3):352-358. doi: 10.1007/s00393-024-01543-6. Epub 2024 Jul 1. PMID 38953936